CLINICAL TRIAL: NCT02231736
Title: Incidence of Chromosomal Damage in Type 2 Diabetes Patients
Brief Title: Chromosomal Damage in Type 2 Diabetes Patients (MIKRODIAB)
Acronym: MIKRODIAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Karl-Heinz Wagner, Director Research Platform Active Ageing, University of Vienna
Other Study IDs: UNIVIE-549-1
Record Dates: First submitted 2014-07-22; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes; Cancer
Keywords: Type 2 Diabetes; Chromosomal damage; Micronuclei; DNA damage; HbA1c; Comet Assay; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 2 diabetes, HbA1c>7.5
- Type 2 diabetes, HbA1c<7.5

SUMMARY:
The purpose of the study is to determine whether glycemic control (HbA1c) is linked to chromosomal damage in type 2 Diabetes patients

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes (T2DM)
* Sex: female
* Age: > 30years
* Medication: oral anti-diabetics and/or Insulin therapy
* Constant nutritional behavior, constant physical activity, constant weight for the last 4 weeks
* Non-smoking for at least 1 year

Exclusion Criteria:

* Patients with type 1 DM
* Age: < 30years
* Pregnant or lactating women
* Participation in another clinical trial
* Change of medication in regard to metabolic parameters within the last 4 weeks
* Significant cardiovascular damage with NYHA > III
* Liver disease with three-times higher transaminase values
* Chronic kidney disease with serum creatinine > 2 mg/dl
* Dialysis
* HIV positive
* History of chronic alcohol abuse in the last two years
* History of cancer, stroke, organ transplantation
* Male

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes patients, female,
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
The quality of HbA1c influences micronuclei formation in binucleated cells | Baseline
  In this cross-sectional study the micronuclei formation in binucleated lymphocytes (Number of micronuclei/1000 binucleated cells) is compared between a low (HbA1c<7.5%) and a high (HbA1c>7.5%) glycemic group

SECONDARY OUTCOMES:
Type 2 diabetes duration of the subjects influences chromosomal damage | Baseline
  The micronuclei formation in binucleated lymphocytes (Number of micronuclei/1000 binucleated cells) is associated with the duration of the Typ 2 diabetes disease.

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Wagner, PhD, Principal Investigator — UNIVIE
Locations (1):
- University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Milic M, Ceppi M, Bruzzone M, Azqueta A, Brunborg G, Godschalk R, Koppen G, Langie S, Moller P, Teixeira JP, Alija A, Anderson D, Andrade V, Andreoli C, Asllani F, Bangkoglu EE, Barancokova M, Basaran N, Boutet-Robinet E, Buschini A, Cavallo D, Costa Pereira C, Costa C, Costa S, Da Silva J, Del Bo' C, Dimitrijevic Sreckovic V, Djelic N, Dobrzynska M, Durackova Z, Dvorakova M, Gajski G, Galati S, Garcia Lima O, Giovannelli L, Goroshinskaya IA, Grindel A, Gutzkow KB, Hernandez A, Hernandez C, Holven KB, Ibero-Baraibar I, Ottestad I, Kadioglu E, Kazimirova A, Kuznetsova E, Ladeira C, Laffon B, Lamonaca P, Lebailly P, Louro H, Mandina Cardoso T, Marcon F, Marcos R, Moretti M, Moretti S, Najafzadeh M, Nemeth Z, Neri M, Novotna B, Orlow I, Paduchova Z, Pastor S, Perdry H, Spremo-Potparevic B, Ramadhani D, Riso P, Rohr P, Rojas E, Rossner P, Safar A, Sardas S, Silva MJ, Sirota N, Smolkova B, Staruchova M, Stetina R, Stopper H, Surikova EI, Ulven SM, Ursini CL, Valdiglesias V, Valverde M, Vodicka P, Volkovova K, Wagner KH, Zivkovic L, Dusinska M, Collins AR, Bonassi S. The hCOMET project: International database comparison of results with the comet assay in human biomonitoring. Baseline frequency of DNA damage and effect of main confounders. Mutat Res Rev Mutat Res. 2021 Jan-Jun;787:108371. doi: 10.1016/j.mrrev.2021.108371. Epub 2021 Feb 6. PMID 34083035